CLINICAL TRIAL: NCT02288585
Title: The Effect of a Low-fat Spread Enriched With Plant Sterol Esters on the Blood Lipid Profile of Subjects With Established Type 2 Diabetes Mellitus and Subjects at High Risk of Developing Type 2 Diabetes
Brief Title: The Effect of Plant Sterols on the Blood Lipid Profile of Subjects With and at High Risk of Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Commonwealth Scientific and Industrial Research Organisation, Australia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FDS-SCC-1552
Record Dates: First submitted 2014-11-04; First posted 2014-11-11 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Vascular Diseases; Hypercholesterolemia; Diabetes Mellitus
Keywords: plant sterols; blood lipids
MeSH Terms: conditions — Vascular Diseases; Hypercholesterolemia; Diabetes Mellitus | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plant sterols (Active Comparator): Plant sterols
  Interventions: Dietary Supplement: Plant sterols
- Placebo product (Placebo Comparator): Placebo product
  Interventions: Dietary Supplement: Placebo product

INTERVENTIONS:
Dietary Supplement: Plant sterols — Plant sterols
  Arms: Plant sterols
Dietary Supplement: Placebo product — Placebo product
  Arms: Placebo product

SUMMARY:
Double-blind, randomised, placebo-controlled, parallel group study with two intervention arms. The study will be conducted in 150 subjects and the primary objective is to show a fasting LDL-cholesterol and triglyceride lowering effect of plant sterols in subjects with established type 2 diabetes mellitus and subjects at high risk of developing type 2 diabetes.

DETAILED DESCRIPTION:
The main aim of the study is to investigate the effect of plant sterols on fasting triglycerides and LDL-cholesterol concentrations.

This study also aims to study the effect of plant sterols on fasting total cholesterol, HDL-cholesterol concentrations and Lipoprotein (a). Furthermore the effects of plant sterols on fasting blood glucose and insulin will be explored. At last, in a sub-group, at end of intervention the acute, chronic and acute upon chronic effect of plant sterols on postprandial blood lipids, glucose and insulin responses during a mixed meal challenge rich in fat and carbohydrates will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Triglycerides >150 mg/dL or 1.74 mmol/L
* LDL-cholesterol: Subjects at high risk for developing T2DM: 115-190 mg/dL or 2.95-4.94 mmol/L. Subjects with established T2DM that are on statins: 85-190 mg/dL or 2.15-4.94 mmol/L.
* HbA1c: Subjects at high risk for developing T2DM: <6.50% or ≥ 48 mmol/mol. Subjects with established T2DM: ≤ 8.5% or ≤ 69 mmol/mol.
* BMI > 20.0 kg/m2.

Exclusion Criteria:

* Recently (within 1 year) diagnosed with cardiovascular event(s) (stroke, TIA, angina, myocardial infarction, heart failure), systemic inflammatory conditions
* Use of over-the-counter and prescribed medication which may interfere with study measurements (i.e. ezetimibe, fibrates and Niacin), to be judged by the principal investigator.
* Currently smoking or being a non-smoker for less than 6 months and reported use of any nicotine containing products in the 6 months prior to screening and/or during the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in TG concentrations | At baseline (after 2 weeks run-in period) and after 6 weeks intervention
Change in LDL-C | At baseline (after 2 weeks run-in period) and after 6 weeks intervention

SECONDARY OUTCOMES:
Change in blood lipids | At baseline (after 2 weeks run-in period) and after 6 weeks intervention

OTHER OUTCOMES:
Change in blood glucose | At baseline (after 2 weeks run-in period) and after 6 weeks intervention
Change in insulin | At baseline (after 2 weeks run-in period) and after 6 weeks intervention
Acute, chronic and acute upon chronic effect on postprandial lipids, glucose and insulin | At the end of intervention (after 6 weeks)
  In a sub-group (n=48) of the population
Change in Advanced Glycation End products (AGEs) | At baseline (after 2 weeks run-in period) and after 6 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Manny Noakes, Principal Investigator — Commonwealth Scientific and Industrial Research Organisation, Australia
Locations (2):
- Australia (2):
  - CSIRO, Adelaide
  - CSIRO, North Ryde, Sydney

REFERENCES:
- [Derived] Trautwein EA, Koppenol WP, de Jong A, Hiemstra H, Vermeer MA, Noakes M, Luscombe-Marsh ND. Plant sterols lower LDL-cholesterol and triglycerides in dyslipidemic individuals with or at risk of developing type 2 diabetes; a randomized, double-blind, placebo-controlled study. Nutr Diabetes. 2018 May 25;8(1):30. doi: 10.1038/s41387-018-0039-8. PMID 29795368